CLINICAL TRIAL: NCT05299528
Title: A Clinician-Focused Nudging Intervention to Optimize Post-Surgical Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Daniel Larach, Asst Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 220508; 5P30AG024968-18 (NIH)
Record Dates: First submitted 2022-03-17; First posted 2022-03-29 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Opioid Prescribing; Surgical Procedure, Unspecified

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Feedback (Experimental): On approximately study day 97, surgeon participants will receive procedure-specific direct feedback through electronic and written communication, on patients' opioid consumption-to-prescription ratio. Surgeon participants who perform more than 1 of the specified procedures will receive nudging communications for each individual procedure.
  Interventions: Behavioral: Direct Feedback
- No Direct Feedback (No Intervention): Surgeon participants randomized to No Direct Feedback will not be contacted directly at any time in the study and will not receive feedback about patients' opioid consumption-to-prescription ratio.

INTERVENTIONS:
Behavioral: Direct Feedback — Procedure-specific direct feedback will be provided to surgeon participants through electronic and written communication, on patients' opioid consumption-to-prescription ratio. Surgeon participants who perform more than 1 of the specified procedures will receive nudging communications for each individual procedure.
  Arms: Direct Feedback

SUMMARY:
This is a pilot single site randomized controlled trial to assess the feasibility and acceptability of a nudging intervention providing surgeons with procedure-specific feedback regarding patients' postoperative opioid prescription-to-consumption ratio in individuals 18 years of age and older.

DETAILED DESCRIPTION:
The trial will randomize surgeons to either intervention (direct feedback) or control (no direct feedback) arms. Surgeons who frequently performing specific elective general, gynecologic, orthopedic, and neurologic surgeries at Vanderbilt University Medical Center will be identified during a 30-day study lead-in period. Then, patients aged at least 18 years undergoing these surgeries at VUMC during study days 1-60 will be contacted by telephone 14 days postoperatively (study days 15-74) and asked to perform an opioid pill count; they will also be asked about opioid refills, satisfaction with analgesia, emergency room visits or hospitalizations for pain, and opioid misuse. The electronic medical record will be also queried for the size of the initial postoperative opioid prescription as well as evidence of any refills for each enrolled subject. Following the first block of surgeries and associated patient follow-up (study days 1-74), data will be analyzed and then surgeons will be randomized in a 1:1 ratio to the intervention or control arms. Randomization will be stratified by both surgical specialty and by mean opioid prescription size during the initial block of surgeries. After study day 97, surgeons in the intervention arm will be provided procedure-specific direct feedback on opioid prescribing and consumption for their patients who had surgery during days 1-60.

After this intervention, the trial will assess pre-post change in opioid prescription size (measured in oral morphine equivalents) from baseline between the two groups for surgeries performed during days 108-167.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Aged greater or equal to 18 years
* Undergoing specified elective general, gynecologic, orthopedic, and neurological surgeries at VUMC during the specified study periods (days 1-60 for the initial patient group; days 105-164 for the follow-up patient group)

  * General: laparoscopic or open cholecystectomy, laparoscopic or open appendectomy
  * Gynecologic: abdominal hysterectomy, laparoscopic/robotic hysterectomy, vaginal hysterectomy, anterior repair/colporrhaphy, posterior repair/colporrhaphy, tension-free vaginal tape procedure, sacrospinous ligament suspension sacrocolpopexy
  * Orthopedic: total knee arthroplasty, total hip arthroplasty, total shoulder arthroplasty, 1- or 2-level spinal laminectomy (without fusion)
  * Neurological: 1- or 2-level spinal laminectomy (without fusion)
* Provided postoperative opioid prescription (verified in VUMC electronic medical record (EMR)
* Able to understand study procedures and participate in the pill count and telephone/electronic interview process in English or Spanish
* Able to provide informed consent

Exclusion Criteria for Patients:

* Opioid prescription filled (per VUMC EMR and patient self report) between 3 months and 7 days prior to surgery
* Primary reason for surgery as assessed by chart review is cancer-related
* Surgery is a repeat/revision surgery (e.g., revision total knee arthroplasty)
* Patient has been inpatient for >3 days postoperatively prior to receiving post-discharge prescription
* Vulnerable populations: current pregnancy, prisoners
* Prior participation in the study (e.g., a patient included in the initial patient group will not be recontacted for the follow-up patient group)

Inclusion Criteria for Surgeon Participants

-General, gynecologic, orthopedic, or neurological surgeon at VUMC during the study period performing any of the surgeries listed below

* General: laparoscopic or open cholecystectomy, laparoscopic or open appendectomy
* Gynecologic: abdominal hysterectomy, laparoscopic/robotic hysterectomy, vaginal hysterectomy, anterior repair/colporrhaphy, posterior repair/colporrhaphy, tension- free vaginal tape procedure, sacrospinous ligament suspension sacrocolpopexy
* Orthopedic: total knee arthroplasty, total hip arthroplasty, total shoulder arthroplasty, 1- or 2-level spinal laminectomy (without fusion)
* Neurological: 1- or 2-level spinal laminectomy (without fusion)

Exclusion Criteria for Surgeon Participants - None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Larach, MD, MSTR, MA, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Surgeon recruitment began on 12/01/2022 and ended on 12/31/2022. Patient recruitment for Phase 1 began on 1/15/2023 and continued through 3/15/2023. Phase 2 recruitment began on 5/22/2023 and ended on 6/30/2023.
Pre-assignment Details: 94 surgeons were identified as potential participants in the study. 27 did not meet eligibility criteria. 20 did not agree to participate. 47 were consented and enrolled into the study. 12 surgeons met criteria to be randomized following Phase 1 Patient Recruitment period.
  Patients who underwent surgery performed by a surgeon who received the nudge intervention were patients who were analyzed only for safety and were not included in other groups. There was a waiver of consent for this group.
Groups:
- Non-Randomized Surgeons Recruited: Surgeons were recruitment on Days -30 through 0. Surgeons who agreed to participate were consented and their patients were screened for Phase 1
- Phase 1 Patient Participants: Patients who were enrolled into Phase 1 of the study prior to randomization of the surgeons to receive the nudge intervention.
- Phase 2 Patient Participants in the Direct Feedback Group: Patients who underwent surgery with a surgeon who was randomized to the direct feedback intervention
- Phase 2 Patient Participants in the No Direct Feedback Group: Patients who underwent surgery with a surgeon who was randomized to the No Direct Feedback Group
- Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention: Patients who underwent surgery performed by a surgeon who received the nudge intervention for 30 days after the intervention
Period: Surgeon Recruitment
Arm/Group | Non-Randomized Surgeons Recruited | Phase 1 Patient Participants | Direct Feedback | No Direct Feedback | Phase 2 Patient Participants in the Direct Feedback Group | Phase 2 Patient Participants in the No Direct Feedback Group | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention
Started (In this initial recruitment phase, only surgeons were recruited.) | 35 | 0 | 6 | 6 | 0 | 0 | 0
Surgeon Recruitment | 35 | 0 | 6 | 6 | 0 | 0 | 0
Completed | 35 | 0 | 6 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 1 Patient Recruitment
Arm/Group | Non-Randomized Surgeons Recruited | Phase 1 Patient Participants | Direct Feedback | No Direct Feedback | Phase 2 Patient Participants in the Direct Feedback Group | Phase 2 Patient Participants in the No Direct Feedback Group | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention
Started (During Phase 1, patient participants from the surgeons enrolled in the surgeon recruitment phase were enrolled in the study) | 0 (Surgeons were not participants in phase 1.) | 135 (Patient participants were not part of the previous period.) | 0 | 0 | 0 | 0 | 0
Completed | 0 | 131 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — 4 patient participants were not eligible after consent. | 0 | 4 | 0 | 0 | 0 | 0 | 0
Period: Surgeon Randomization
Arm/Group | Non-Randomized Surgeons Recruited | Phase 1 Patient Participants | Direct Feedback | No Direct Feedback | Phase 2 Patient Participants in the Direct Feedback Group | Phase 2 Patient Participants in the No Direct Feedback Group | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention
Started (35 surgeons who did not have at least 3 patients who had specified surgeries during phase 1 were not randomized) | 0 (Surgeons were not participants in Phase 1.) | 0 (Patient participants were not part of the previous period.) | 6 (Surgeons were not participants in Phase I.) | 6 (Surgeons were not participants in Phase I.) | 0 | 0 | 0
Completed | 0 | 0 | 6 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2 Patient Recruitment
Arm/Group | Non-Randomized Surgeons Recruited | Phase 1 Patient Participants | Direct Feedback | No Direct Feedback | Phase 2 Patient Participants in the Direct Feedback Group | Phase 2 Patient Participants in the No Direct Feedback Group | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention
Started (During Phase 2, patient participants from the surgeons who were randomized to receive the Direct or No Direct Feedback Intervention were enrolled in the study. The 58 patient participants in this period are not included in the 135 patient participants enrolled in Phase 1 Patient Recruitment.) | 0 (Surgeons were not participants in Phase 2.) | 0 | 0 (Surgeons were not participants in Phase 2.) | 0 (Surgeons were not participants in Phase 2.) | 27 (Patient participants were not part of the previous period.) | 31 (Patient participants were not part of the previous period.) | 225 (These patients were not participants in the previous period.)
Completed | 0 | 0 | 0 | 0 | 27 | 30 | 225
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant was determined to be ineligible after consent | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Surgeon Follow-up
Arm/Group | Non-Randomized Surgeons Recruited | Phase 1 Patient Participants | Direct Feedback | No Direct Feedback | Phase 2 Patient Participants in the Direct Feedback Group | Phase 2 Patient Participants in the No Direct Feedback Group | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention
Started | 0 | 0 | 6 (Surgeons were not participants in the previous period.) | 6 (Surgeons were not participants in the previous period.) | 0 (Patient participants were not part of this period.) | 0 (Patient participants were not part of this period.) | 0 (These patients were not participants in this period.)
Completed | 0 | 0 | 5 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-randomized Surgeons Recruited: Non-randomized surgeons recruited to participate in the study
- Phase 2 Patient Participants in the No Direct Feedback Group: Patients who underwent surgery with a surgeon who was randomized to the no direct feedback intervention
- Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention: Patients who underwent surgery performed by a surgeon who received the nudge intervention for 30 days after the intervention. Does not include Phase 2 patient participants. Adverse events were assessed at post op days 10 and 30.
- Total: Total of all reporting groups
Arm/Group | Non-randomized Surgeons Recruited | Phase 1 Patient Participants | Direct Feedback | No Direct Feedback | Phase 2 Patient Participants in the Direct Feedback Group | Phase 2 Patient Participants in the No Direct Feedback Group | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention | Total
Number analyzed (Participants) | 35 | 135 | 6 | 6 | 27 | 31 | 225 | 465
Age, Categorical [Count of Participants; unit: Participants] — Population: The group "Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention" did not have age, sex, race or ethnicity data collected.
  Participants
    number analyzed (Participants) | 35 | 135 | 6 | 6 | 27 | 31 | 0 | 240
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 35 | 76 | 5 | 4 | 20 | 21 | 0 | 161
    >=65 years | 0 | 59 | 1 | 2 | 7 | 10 | 0 | 79
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Patients in the arm "Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention" did not have age, sex, race or ethnicity data collected.
  Participants
    number analyzed (Participants) | 35 | 135 | 6 | 6 | 27 | 31 | 0 | 240
    Female | 12 | 87 | 1 | 1 | 20 | 21 | 0 | 142
    Male | 23 | 48 | 5 | 5 | 7 | 10 | 0 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race/Ethnicity data was not collected for the surgeon participants. Patients in the arm "Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention" did not have age, sex, race or ethnicity data collected.
  Participants
    number analyzed (Participants) | 0 | 135 | 0 | 0 | 27 | 31 | 0 | 193
    Hispanic or Latino |  | 4 |  |  | 1 | 0 | 0 | 5
    Not Hispanic or Latino |  | 100 |  |  | 24 | 30 | 0 | 154
    Unknown or Not Reported |  | 31 |  |  | 2 | 1 | 0 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race/Ethnicity data was not collected for the surgeon participants
  Participants
    number analyzed (Participants) | 0 | 135 | 0 | 0 | 27 | 31 | 0 | 193
    American Indian or Alaska Native |  | 1 |  |  | 1 | 0 | 0 | 2
    Asian |  | 0 |  |  | 0 | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander |  | 0 |  |  | 0 | 0 | 0 | 0
    Black or African American |  | 12 |  |  | 6 | 4 | 0 | 22
    White |  | 114 |  |  | 19 | 26 | 0 | 159
    More than one race |  | 2 |  |  | 1 | 0 | 0 | 3
    Unknown or Not Reported |  | 6 |  |  | 0 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 35 | 135 | 6 | 6 | 27 | 31 | 225 | 240

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Surgeons Approached Who Agree to Participate
Description: Feasibility outcome: Percentage of surgeons approached who agree to participate in study
Time Frame: At consent (study days -30 to 0)
Population: Total number of potentially eligible surgeons who were eligible
Measure: Count of Participants; unit: Participants
Groups:
- Surgeon Recruitment: Surgeons were recruitment on Days -30 through 0. Surgeons who agreed to participate were consented and their patients were screened for Phase 1
Arm/Group | Surgeon Recruitment
Number analyzed (Participants) | 94
Participants | 47

2. Primary Outcome: Percentage of Patients Contacted Who Agree to Participate in Study
Description: Feasibility outcome: Percentage of patients contacted who agree to participate in study
Time Frame: At consent (single time during study days 15-74 (group 1) or 122-181 (group 2))
Population: Total number of potentially eligible patients who were contacted about participation.
  Patients who underwent surgery performed by a surgeon who received the nudge intervention were patients who were analyzed only for safety. They were not contacted about the study, and were not included in the primary outcome analysis. This group was enrolled with a waiver of consent.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Patient Participants | Phase 2 Patient Participants in the Direct Feedback Group | Phase 2 Patient Participants in the No Direct Feedback Group
Number analyzed (Participants) | 228 | 42 | 66
Participants | 135 | 27 | 31

3. Primary Outcome: Surgeon-reported Acceptability of Intervention
Description: Acceptability outcome: Surgeon-reported acceptability of intervention as measured by a "yes" response to the question "Would you find receiving such feedback on your patients' opioid consumption acceptable?"
Time Frame: Post intervention (once on study day 181)
Population: One surgeon randomized to the direct feedback group did not complete the post-study survey
Measure: Count of Participants; unit: Participants
Arm/Group | Direct Feedback | No Direct Feedback
Number analyzed (Participants) | 5 | 6
Participants | 5 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected on patients who had surgery following the surgeon nudge intervention on Day 97
Description: Adverse events were not monitored in surgeon participants or Phase 1 patient participants.
Arm/Group | Phase 2 Patient Participants in the Direct Feedback Group | Phase 2 Patient Participants in the No Direct Feedback Group | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/31 | 0/225
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/31 | 5/225
Other Adverse Events (participants affected / at risk) | 2/27 | 1/31 | 5/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 Patient Participants in the Direct Feedback Group (N=27) | Phase 2 Patient Participants in the No Direct Feedback Group (N=31) | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention (N=225)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — Intractable vomiting that required inpatient hospitalization for IV fluids and medication
Abdominal pain (Surgical and medical procedures) | 0 (0) | 0 (0) | 3 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Clostridioides difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 2 Patient Participants in the Direct Feedback Group (N=27) | Phase 2 Patient Participants in the No Direct Feedback Group (N=31) | Patients Who Underwent Surgery Performed by a Surgeon Who Received the Nudge Intervention (N=225)
Pain (General disorders) | 1 (1) | 1 (1) | 2 (2) — Post-operative pain following surgery
diverticulosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — GI bleeding secondary to diverticulosis
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
* Not powered for efficacy
* Cohort was mostly non-Hispanic white
* Participants self-reported pill count
* Surgeons did not remember the nudge

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT05299528/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT05299528/ICF_000.pdf